CLINICAL TRIAL: NCT02960672
Title: Sequential Changes of Serum KL-6 Predict Progression in Interstitial Lung Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Ying Jiang, Director, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: gyfyy
Record Dates: First submitted 2016-10-27; First posted 2016-11-10 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Interstitial Lung Disease, Desquamative
Keywords: KL-6; disease progression; predict; biomarkers; MMP-7
MeSH Terms: conditions — Interstitial Pneumonitis, Desquamative, Familial; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood biomarkers
Oversight: Data Monitoring Committee: No

SUMMARY:
Interstitial lung disease is a chronic progressive fibrosis lung disease that with a highly variable clinical process.thence it is significant for the patient to search a convenient and accurate prediction method. The objective of this study was to determine whether peripheral blood biomarkers can predict disease .

DETAILED DESCRIPTION:
The median follow-up period was 12 months, each patient received 4 or 5 follow-ups in our center, 336 person-times in study enrollment totally. The patients with interstitial lung disease had significantly higher serum baseline KL-6 and MMP-7 levels compared with healthy control.They divided into progressive group and non-progressive group according to disease change. Serum KL-6 and MMP-7 levels were elevated in patients if disease progression, but baseline level of biomarkers in progressive group were not significant higher compare with non-progressive group .Binary logistic regression showed △KL-6 and △MMP-7 were significant predictors for disease progression. Multivariate Cox analysis showed KL-6 and MMP-7 were significantly associated with survival along with other variables.

The serum levels of KL-6 and MMP-7 were elevated in the individuals with interstitial lung disease compared with healthy controls. The rate of poor prognosis and mortality more associated with the variability increased biomarker concentrations，rather than the baseline concentration.Therefore，Serial measurements of biomarkers contribute to the disease monitoring in clinical management.

ELIGIBILITY:
Inclusion Criteriar:

* Clinical diagnosis of interstitial lung disease

Exclusion Criteria:

* Diagnosise of interstitial lung disease acute excerbation
* Combined pulmonary embolism, pulmonary edema, pulmonary tuberculosis, and peumonias

Ages: 40 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects with a diagnosis of idiopathic interstitial pneumonias made in accordance with the American Thoracic Society (ATS)/European Respiratory Society (ERS) consensus classification
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-03; Primary Completion 2016-10 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Sequential Changes of Serum KL-6 Predict Progression in Interstitial Lung Disease | 3 years
  Serum samples were prospectively collected from 70 patients including baseline, 1 month, 2 months, 6 months and 12 months, which were tested for a panel of Krebs van den Lungen-6 antigen (KL-6), by latex agglutination test.We have demonstrated that an increase in serum KL-6 levels, but not the level at any one point in time, predicts poor prognosis.

SECONDARY OUTCOMES:
Sequential Changes of Serum MMP-7 Predict Progression in Interstitial Lung Disease | 3 years
  Serum samples were prospectively collected from 70 patients including baseline, 1 month, 2 months, 6 months and 12 months, which were tested for a panel of matrix metalloproteinase-7 (MMP-7), by ELISA-based.We have demonstrated that an increase in serum MMP-7 levels, but not the level at any one point in time, predicts poor prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Ying Jiang, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No